CLINICAL TRIAL: NCT04265339
Title: The Interplay Between Addiction to Tobacco Smoking and Sleep Quality Among Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Max Stern Academic College Of Emek Yezreel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1497/17
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Tobacco Dependence
Keywords: Sleep; Tobacco Smoking; Smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Three study groups: Smokers, non-smokers and smoking cessation group.
Who Masked: Outcomes Assessor
Masking Description: The data analysis will be conducted without knowledge of the group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- None smokers (No Intervention): 50 participants who are non-smokers
- Smoking Cessation (Experimental): 50 smokers who quit smoking
  Interventions: Other: Smoking cessation
- Active smokers (No Intervention): 50 smokers who continue smoking

INTERVENTIONS:
Other: Smoking cessation — Participants are required to quit smoking
  Arms: Smoking Cessation

SUMMARY:
Tobacco smoking is a major health problem, leading to considerable morbidity and mortality due to cancer, impaired pulmonary function, and cardiovascular diseases. Chronic nicotine consumption related to smoking may affect pulmonary function and can cause neuronal alterations leading to increased emotional distress and decreased cognitive functioning, especially when the smoker attempts to quit. These may explain the huge difficulty in quitting and the dependence on cigarettes as a means of maintaining emotional balance. The possibility that reduced sleep quality is a major negative outcome that contributes to nicotine addiction has been largely overlooked. Several studies have shown that smoking and smoking cessation disrupt sleep quality; however, the vast majority of these studies were based on subjective reports. Moreover, it is not clear to what degree disrupted sleep quality among smokers may be related to reduced pulmonary function, and to what degree reduced sleep quality contributes to the emotional cognitive distress of active and abstinent smokers and to their urge to smoke. The main hypothesis of this proposal is that smoking and early phases of smoking cessation will be associated with reduced sleep quality. This poor sleep quality will be associated with emotional and cognitive symptoms and difficulty in abstaining from tobacco smoking. Successful abstinence from smoking over time will lead to normalization of the quality of sleep.

Experiments to investigate this hypothesis will be conducted on healthy young adults addressing the following specific aims: 1) To examine physiological and psychological factors predicting reduced quality of sleep among smokers, including: poor pulmonary function, the degree of nicotine dependence, altered regulation of stress systems (HPA axis and the sympathetic nervous system), and emotional distress (anxiety and depression); 2) To explore the impact of smoking cessation on sleep quality and related symptoms. Specifically, whether smoking cessation induces fragmented sleep and poor sleep quality, and whether the diminished sleep quality can predict the magnitude of emotional and cognitive symptoms; 3) To examine whether poor sleep (before and during abstinence) can predict the level of the urge to smoke and smoking relapse among abstinent smokers; 4) To explore whether sleep quality ultimately improves following prolonged abstinence from smoking. Addressing these aims, nonsmokers and smokers will be examined before and during smoking abstinence on the following measures: quality of sleep via actigraphy and polysomnography (PSG), pulmonary function test, biological markers of stress (cortisol and α-amylase) and smoking (i.e., cotinine, the main metabolite of nicotine), and emotional and cognitive functioning via psychometric tests.

Results of this study will provide novel insight on the role of sleep in nicotine addiction. Experiments will show how reduced quality of sleep may result from chronic smoking and interfere with attempts to quit smoking. Also, the experiment will shed light on the interrelated physiological and psychological mechanisms that mediate the interplay between smoking addiction and sleep. The research will utilize a variety of powerful methods and an interdisciplinary collaboration of experts in the fields of sleep, addiction, and pulmonary medicine. It is anticipated that the results will contribute substantially to our knowledge of smoking addiction and may promote the development of effective therapeutic interventions to this major public health problem.

DETAILED DESCRIPTION:
Scientific background Tobacco smoking is a major health problem, leading to considerable morbidity and mortality due to cancer, pulmonary illnesses, and cardiovascular diseases (Taghizadeh, Vonk & Boezen, 2016). The main psychoactive and addictive substance in tobacco is nicotine (Zaparoli & Galduroz, 2012). Nicotine addiction is a complex phenomenon that involves both physical and psychological dependence (Cohrs et al., 2014), which causes not only difficulty in quitting but also a strong tendency to return to smoking after having quit for a long time) Zaniewska, Przegalinski & Fillip, 2009).

A common theoretical model of addiction (Koob & Volkow, 2016) holds that the transition from occasional smoking to addiction involves an upregulation of neurobiological stress systems. Consequently, even a brief period of abstinence from smoking, leading to reduced concentration of nicotine in the body, induces both emotional withdrawal symptoms (anxiety, restlessness, irritability, anhedonia) and cognitive withdrawal symptoms (diminished memory and attention) that may in turn produce a compulsive urge to smoke again, in order to ease the unpleasant sensations (Koob & Volkow, 2016). Although some studies suggest reduced quality of sleep is also among the consequences of smoking and smoking cessation (Cohrs et al., 2014; Colrain, Trinder & Swan, 2004) this issue was not fully explored, and the contribution of the reduced quality of sleep to negative emotional situations and to the motivation to smoke is unclear.

Smoking and sleep. Smokers report more sleep disturbances such as insomnia (i.e., a variety of complaints reflecting dissatisfaction with the ability to initiate and maintain sleep, along with a significant reduction in total sleep time followed by daytime sleepiness) (Kaneita et al., 2005; Phillips & Danner, 1995), and a correlation was found between the level of addiction to cigarettes and reduced quality of sleep (Palmer, Harrison & Hiorns, 1980; Patten et al., 2000). A deleterious effect of smoking on the quality of sleep could partially result from disturbed pulmonary function (Simon-Tuval et al., 2011). Indeed, heavy smokers are at high risk for Chronic Obstructive Pulmonary Disease (COPD) (Tarasiuk et al., 2006), which causes disturbed sleep leading to reduced quality of life (Scharf et al., 2011; Won & Kryger, 2014). Moreover, even in young, seemingly healthy, moderate smokers there is a clear reduction in pulmonary function, and a negative correlation was found in healthy adults between pulmonary functioning and sleep quality (Phillips et al., 1989). However, this factor could not solely explain the relationship between smoking and quality of sleep, as studies have shown an increased number of awakenings in the course of the night during early phases of smoking cessation (Hatsukami, Hughes & Pickens, 1985; Hatsukami et al., 1988).

The reliability of subjective sleep measures is not unequivocal and needs support from objective measurements (Pillar, Malhotra & Lavie, 2000). To date, only a handful of studies compared the sleep architecture of active and quitting smokers to that of nonsmokers using polysomnographic (PSG) tests (consisting of brain wave, muscle tension, eye movement, and other measurements). These studies confirmed the deleterious effects of smoking and smoking cessation on the quality of sleep. Zhang and colleagues (2006) found that compared to nonsmokers, the sleep of smokers was characterized by shorter duration, longer time to reach (rapid eye movement) REM sleep, longer time spent in light sleep (stage 1), less time spent in deep sleep (stages 3 and 4, slow-wave sleep-SWS), and lower sleep efficiency (percentage of actual sleep time of the total time spent in bed). Similarly, sleep duration among smokers was shorter than among nonsmokers (Jaehne et al., 2012). Likewise, PSG tests conducted on individuals undertaking smoking cessation demonstrated increases in the number of awakenings at night (Prosise et al., 1994), shortening of REM latency, shortening of SWS sleep duration, and extension of the phases of light sleep (stages 1 and 2) (Moreno-Coutiño, Calderón-Ezquerro & Drucker-Colín, 2007; Wetter et al., 2000), all indications of reduced quality of sleep. Yet, these PSG studies also had limitations as they were usually conducted on a small number of patients on a single night, under the artificial conditions of sleep laboratories.

Quality of sleep, stress, and addiction to smoking. It is well accepted that sleep plays a vital role in health as well as behavioral and emotional stability (Scharf et al., 2010; Tarasiuk et al., 2005). Those who suffer from poor sleep quality exhibit higher rates of psychological stress, depression, and various anxiety symptoms than the general population (Fernández-Mendoza et al., 2009; Ohayon, 2005). The tendency toward poor sleep quality among smokers and quitters, and the correlation between proper sleep and behavioral and emotional stability raise the hypothesis that the impairment in sleep quality among smokers and quitters affects their psychological functioning and their smoking behavior. The few studies that investigated this issue demonstrated that abstaining from cigarette smoking for 48 hours increased the subsequent rate of smoking (Hamidovic& de Wit, 2009), and that sleep disruptions during withdrawal have a negative effect on the success of smoking cessation (Jaehne et al., 2009; Persico, 1992). These findings seem to integrate well into the aforementioned theoretical model, which holds that exposure to nicotine leads to the development of aversive psychological symptoms when the bodily nicotine concentration drops, which leads to a compulsive urge to smoke to alleviate these unpleasant sensations (Cohen & George, 2013).

A variety of findings suggest that these aversive psychological symptoms are due to an increase in the activity of neurobiological systems that regulate stress responses (Cohen & George, 2013). Stress responses are regulated by two key neuroendocrinological systems: the sympathetic nervous system and the HPA (hypothalamus-pituitary-adrenocortical) axis. The sympathetic system is responsible for increasing the level of arousal in situations of danger and acute stress. It involves mainly the secretion of adrenaline by the adrenal gland. Studies indicate that level of the α-amylase enzyme in the saliva is an indirect but reliable measure of sympathetic activity (Rohleder et al., 1994). It has been demonstrated that the α-amylase levels before and after smoking cessation predicted the measure of success in persisting with abstinence from smoking over time (Duskova et al., 2010). The HPA system regulates physiological reactions related to coping with ongoing stressors. Specifically, it induces secretion of the Corticotrophin Releasing Hormone (CRH) from the paraventricular nucleus, located in the hypothalamus, to the anterior pituitary gland, which in response secretes the AdrenoCorticoTropic Hormone (ACTH) that stimulates the release of cortisol by the adrenal gland (Ma et al., 2011). Cortisol levels in the body generally rise sharply in response to stressors, but in people who are in chronic stress situations, regulation of the HPA system may be disrupted, which is manifested by reduced secretion of cortisol both in the basal situation and in response to stress (Miller, Chen & Zhou, 2007). This sub-regulation may reflect difficulty in coping with stress (Miller, Chen & Zhou, 2007): low levels of cortisol are associated with an increased level of depression (Moraes et al., 2016), aggression (Granger, 1998), and impulsiveness (Blomqvist et al., 2007). Note that while acute exposure to nicotine increases levels of cortisol temporarily (Newhouse et al., 1990; Winternitz & Quillen, 1977), secretion of cortisol in chronic smokers in response to stress is reduced relative to that of nonsmokers (Kirschbaum, Strasburger & Langkrär, 1993; Rohleder & Kirschbaum, 2006). Moreover, studies indicate a decrease in cortisol levels during smoking cessation (Steptoe & Ussher, 2006; Targovnik,1989), which correlates with the intensity of the somatic and emotional withdrawal symptoms and with the level of the urge to smoke (Cohen, al'Absi & Collins, 2004; Targovnik,1989); it also correlates with the level of success in persisting with smoking cessation over time (al'Absi et al.,2004; Frederick et al., 1998). This may be due to the development of sub-regulation by the HPA system, similarly to the situation of those suffering from chronic stress (Richardson et al., 2008), which in turn leads to the sensitization of the mechanisms of stress in the brain, such as increasing the activity of CRH in the limbic system (Vendruscolo et al., 2012). The literature partially supports the possibility that an increase in the activity of neurobiological stress mechanisms (due to chronic exposure to nicotine) contributes to disruption of the quality of sleep. For example, increased sympathetic activity during the day, as reflected in high levels of α-amylase, is highly correlated with insomnia (Nater et al., 2007). However, various studies that have examined the relationship between different measures of cortisol secretion throughout the day and night, and various indices of sleep, produced conflicting results (Elder et al., 2014). Recent studies indicate that cortisol is produced at a higher rate during REM sleep; therefore, prolonged sleep, which includes longer REM sleep, produces higher cortisol levels (Van Lenten & Doane, 2016). Note that whereas an increase in the levels of stress may disrupt sleep, poor sleep quality may in itself cause stress (Fernández-Mendoza et al., 2009; Ohayon, 2005).

In sum, several studies suggest that smoking and, even more so smoking cessation, disrupt sleep, and that the reduced quality of sleep may contribute to the motivation to smoke and reduce the prospects for quitting. However, the number of these studies is relatively small, and many of them are based on subjective reports, whose reliability is not unequivocal. The minority of studies that used objective measurements usually tested a small number of participants, under the artificial conditions of the sleep laboratory. Notably, the quality of sleep can be measured objectively and reliably for extended periods of time in the participants' natural environment using an actigraph device that is worn on the wrist and analyzes movement (Ancoli-Israel et al., 2015; Sadeh et al., 1989). However, actigraphy has not been used thus far for assessing the sleep quality of smokers. Moreover, to date there has been no systematic study of the complex relations between sleep, pulmonary function, stress systems functioning, and smoking as they relate to the development and persistence of tobacco smoking addiction.

We hypothesize that chronic tobacco smoking impairs sleep quality, which in turn enhances the activity of stress mechanisms, and thus induces negative emotional states. The processes that harm sleep quality and the processes that increase responsiveness to stress and negative emotional symptoms thus reciprocally nourish each other and ultimately increase the urge to smoke as a means for stress relief. Our preliminary findings support this hypothesis by demonstrating that active smokers suffer from diminished quality of sleep (assessed by actigraphy and questionnaires), compared to nonsmokers, an effect that was correlated with markers of stress activation, namely levels of cortisol and α-amylase in the participants' saliva.

Research objectives and expected significance

Our research will explore the role of sleep disturbances in tobacco smoking addiction. Based on our preliminary findings and the available literature, the main hypothesis of this proposal is that smoking, and to a greater degree early phases of smoking cessation, will be associated with reduced quality of sleep. The reduced quality of sleep will, in turn, predict the severity of negative symptoms and the extent of difficulty in abstaining from smoking. Successful abstinence from smoking will lead to normalization of sleep. Experiments to investigate this hypothesis will address the following specific aims:

1. To examine physiological and psychological factors predicting reduced quality of sleep among smokers. The goal is to explore the deleterious effects of smoking on sleep quality and to explore whether the reduced sleep quality is predicted by the following factors: poor pulmonary function (FEV1, FEF), degree of nicotine dependence, emotional symptoms (anxiety and depression), and altered regulation of stress systems (HPA axis and the sympathetic nervous system). We expect that, compared to nonsmokers, smokers will exhibit poorer sleep quality. The level of disruption to the quality of sleep will be related to the intensity of nicotine dependence, poor pulmonary functioning, the levels of negative emotionality, sympathetic activation, and deregulation of HPA axis.
2. To explore the impact of smoking cessation on sleep quality and related symptoms. We will examine whether smokers who try to quit experience a worsening sleep quality, and whether this poor sleep quality can predict the magnitude of their stress response (level of cortisol and α-amylase) and the severity of emotional and cognitive symptoms as measured by the psychometric tests.
3. To explore the role of sleep quality on smoking motivation and relapse to smoking. Experiments will determine whether sleep can predict the urge to smoke (in current smokers) and the likelihood of abstinent smokers to relapse.
4. To explore whether prolonged abstinence from nicotine improves sleep quality. The aim here is to examine whether smoking cessation ultimately induces normalization of sleep and related factors, including pulmonary functioning, stress response (level of cortisol and α-amylase), and emotional and cognitive functioning. Smoking abstinence will be verified by measurement of cotinine in the participant's saliva.

Expected Significance. Experiments will show how reduced quality of sleep may result from chronic smoking and interfere with attempts to quit smoking. This study will shed light on the interrelated physiological and psychological mechanisms that mediate the interplay between smoking addiction and sleep, including psychological distress, dysfunctional stress mechanisms, and reduced pulmonary functioning.

The proposed study will utilize a variety of powerful methods and an interdisciplinary collaboration of experts in the fields of sleep, addiction, and respiratory medicine to explore the interplay of sleep and tobacco smoking. Results of this study will provide novel insight on the role of sleep in nicotine addiction. Findings of the proposed research are expected to promote the use of sleep quality enhancement techniques in smoking cessation interventions. Methodology Participants. Participating in the study will be 150 healthy volunteers, men and women, aged 18-30, with no history of mental illness or drug abuse. The number of participants was established by power analysis, based on our preliminary results, with addition of 20% to compensate for possible drop-outs during the study. Fifty participants will be nonsmokers, and the rest regular smokers . Half of the smokers will be with a stated interest in quitting and half with no such interest (non-quitting control). Participants will receive a compensation fee of 400 NIS (roughly 100 US dollars). All procedures used in this study have been approved by Yezreel Valley College (YVC) Institutional Review Board.

Research procedure. Participants will be recruited from the student body of the college and, via advertisement, from the surrounding communities. All study sessions will start between 7:00 AM and 9:00 AM (up to 30 minutes following awakening) either at the YVC Psychobiology Laboratory or in the participant's home.

The study will include 3 groups (N=50): smokers attempting to quit (smoking cessation group, SCG), nonsmokers group (NSG), and a group of smokers not attempting to quit (SNCG). The latter group is needed in order to assure that changes in certain measures following smoking cessation are not due to time-related events that are not related to abstinence from tobacco. The study design includes 4 stages: A) Baseline. B) First week of nicotine cessation. C +D) Follow up tests three months and six months following the initiation of smoking cessation. Note that although the 2 control groups (i.e., the nonsmokers group (NSG) and the group of smokers not attempting to quit (SNCG)) will not undergo smoking cessation, they will be evaluated with the same tests and at the same time points as the smoking cessation group.

Baseline Phase: At the first session, all the participants will be asked to sign a consent form and provide background information. After assessing their smoking status by checking the level of carbon monoxide (CO) in their breath, they will be asked to give a saliva sample (to test the levels of cortisol and α-amylase) by spitting into a test tube (1.5 mL minimum). To further validate the participants' smoking status, the saliva samples will also be used to detect the levels of cotinine, the primary metabolite of nicotine. Participants will be asked to complete a broad spectrum of questionnaires, evaluating their level of anxiety, depression, quality of sleep, and smoking dependence (questionnaires are described in detail below), as well as completing the Cognitive Assessment Battery (CAB), a computerized neurocognitive test designed to assess a large range of cognitive skills related to executive functions. In addition, their pulmonary functioning will be assessed via spirometry. Finally, participants' sleep will be continuously monitored over a 1-week period by a miniature wrist-worn actigraph, and will be recorded during the last two nights of this week by PSG.

Smoking cessation phase: At the end of the baseline week, participants of the smoking cessation study group will begin abstaining from smoking, while participants on the 2 control groups (i.e., the nonsmokers group (NSG) and the group of smokers not attempting to quit (SNCG) will carry on with their regular routine. In the morning of the first day of smoking cessation, all participants will provide saliva samples and complete the same set of questionnaires as in the baseline phase. All participants will then be asked to wear the actigraphy device during the second week as well, and to return to the lab for additional sessions after 48 hours, 72 hours, 5 days, and one week (altogether four times). At each of these sessions, the smoking status of the participants will be assessed by means of the exhalation test, and participants will again be asked to provide a saliva sample, and complete the same set of questionnaires. On the last two nights of this week, participants' sleep will also be recorded by PSG. On the morning of day 7 of abstinence, all participants will also complete (again) the CAB neurocognitive test. Follow up phase: Will be conducted on all participants three months and six months into the smoking cessation process of the smoking abstinence group. At each of these time points, all participants will be summoned for an additional data collection session in which it will be determined who of the smoking abstinence participants relapsed back to smoking. In addition, all participants will again be asked to complete the set of questionnaires and the CAB neurocognitive test. The pulmonary functioning of the participants will again be measured by spirometry and they will be asked to wear the actigraph device for one week. In addition, their sleep will be recorded for two consecutive nights by PSG. Saliva samples collected during the study will destroyed following their ELISA analysis. All participants will be assured of confidentiality and anonymity, and all staff involved in the study will maintain the confidentiality of the study. All material collected will be kept locked in a designated cabinet.

ELIGIBILITY:
Inclusion Criteria:

For the smokers group:

* At least 10 cigarettes a day on average, for the preceding 2 years
* Meeting the criteria for tobacco use disorder laid out in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

For the nonsmokers group:

• Not having smoked more than 5 cigarettes in their lifetime and not at all in the preceding 2 years.

Exclusion Criteria:

* History of mental illness or substance abuse.
* Working on night shifts.
* Pregnancy
* Clinical diagnosis of a sever lung disease, such as Chronic Obstructive Pulmonary Disease (COPD)
* Clinical diagnosis of a severe sleeping disorder, such as sleep apnea, narcolepsy and hypersomnia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Objective Sleep Quality at 6 months | Two weeks at baseline, During first week of smoking cessation, for two weeks 3 month after smoking cessation and for two weeks 6 month after smoking cessation
  Actigraphy
Change from Baseline Sleep Structure at 6 months | Two nights at baseline, one night at the end of the first week of smoking cessation, one night 3 month after smoking cessation and one night 6 month after smoking cessation
  Polysomnography (PSG)
Change from Baseline Subjective Sleep Quality at 6 months | Once at baseline, Once at the end of the first week of smoking cessation,Once 3 month after smoking cessation and Once 6 month after smoking cessation
  The Pittsburgh Sleep Quality Index (PSQI).The questionnaire consists of 19 individual items, generating seven "component" scores: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The component scores are added to yield one "global" score, with a range of 0-21 points, with higher scores indicating more severe sleep difficulties.
Change from Baseline Tobacco Smoking Dependence at 6 months | Once at baseline, Once at the end of the first week of smoking cessation,Once 3 month after smoking cessation and Once 6 month after smoking cessation
  Minnesota Nicotine Withdrawal Scale (MNWS).The questionnaire includes nine items, each describing a specific nicotine withdrawal symptom. Participants indicate the degree of severity with which they experienced each symptom in the preceding 24 hours on a 5-point scale (0-4). The items are averaged for a single severity score (0-4), with a higher score indicating a more severe level of dependence.
Change from Baseline Tobacco Smoking urge at 6 months | Once at baseline, Once at the end of the first week of smoking cessation,Once 3 month after smoking cessation and Once 6 month after smoking cessation
  Brief Questionnaire on Smoking Urges (QSU). consists of 10 items, each a statement referring to the amount of craving for a cigarette at a given point in time. Participants indicate the level of their agreement with each statement on a 7-point Likert scale (1-7). The final score is the sum of all responses (range:10-70), with a higher score indicating a stronger urge to smoke.
Change from Baseline Depressive Symptoms at 6 months | Once at baseline, Once at the end of the first week of smoking cessation, Once 3 month after smoking cessation and Once 6 month after smoking cessation
  Beck's Depression Inventory (BDI-II). Includes 21 items, each consisting of four statements representing increasing levels of severity of a particular depressive symptom. Participants specify which statement best describes their feeling in the preceding week. The scores are added for a final score (0-63), . with a higher score indicating a more severe state of depression.
Change from Baseline State Anxiety at 6 months | Once at baseline, Once at the end of the first week of smoking cessation, Once 3 month after smoking cessation and Once 6 month after smoking cessation
  State-Trait Anxiety Inventory (STAI).The portion of the questionnaire that assesses state anxiety includes 20 items, each a statement relating to the participant's sense of anxiety at that point in time. Participants indicate agreement with each statement on a 4-point scale (1-4). The scores are added for a final score (20-80), with a higher score indicating a more severe state of anxiety.
Change from Baseline Biological Markers of Stress and Tobacco Smoking at 6 months | Once at baseline, Once at the end of the first week of smoking cessation, Once 3 month after smoking cessation and Once 6 month after smoking cessation
  Salivary levels of cortisol, α-amylase, and cotinine
Change from Baseline Exhaled Carbon Monoxide at 6 months | Once at baseline, 4 times during the first week of smoking cessation (day 2, day 3, day 5, day 7), Once 3 month after smoking cessation and Once 6 month after smoking cessation
  Carbon monoxide (CO) exhalation level
Change from Baseline Cognitive Functioning at 6 months | Once at baseline, Once at the end of the first week of smoking cessation,Once 3 month after smoking cessation and Once 6 month after smoking cessation
  Cognitive Assessment Battery (CAB)
Change from Baseline Pulmonary Function as measured by spirometry (the volume and speed of air that can be inhaled and exhaled) at 6 months | Once at baseline, Once at the end of the first week of smoking cessation, Once 3 month after smoking cessation and Once 6 month after smoking cessation
  The parameters measured in spirometry are Vital Capacity (VC), Forced Vital Capacity (FVC), Forced Expiratory Volume (FEV), Forced Expiratory Flow (FEF), and Maximal Voluntary Ventilation (MVV).

CONTACTS AND LOCATIONS:
Locations (1):
- The Max Stern Academic College of Emek Yezreel, Afula, Israel

REFERENCES:
- [Background] al'Absi M, Hatsukami D, Davis GL, Wittmers LE. Prospective examination of effects of smoking abstinence on cortisol and withdrawal symptoms as predictors of early smoking relapse. Drug Alcohol Depend. 2004 Mar 8;73(3):267-78. doi: 10.1016/j.drugalcdep.2003.10.014. PMID 15036549
- [Background] Ancoli-Israel S, Martin JL, Blackwell T, Buenaver L, Liu L, Meltzer LJ, Sadeh A, Spira AP, Taylor DJ. The SBSM Guide to Actigraphy Monitoring: Clinical and Research Applications. Behav Sleep Med. 2015;13 Suppl 1:S4-S38. doi: 10.1080/15402002.2015.1046356. No abstract available. PMID 26273913
- [Background] Blomqvist M, Holmberg K, Lindblad F, Fernell E, Ek U, Dahllof G. Salivary cortisol levels and dental anxiety in children with attention deficit hyperactivity disorder. Eur J Oral Sci. 2007 Feb;115(1):1-6. doi: 10.1111/j.1600-0722.2007.00423.x. PMID 17305710
- [Background] Cohen A, George O. Animal models of nicotine exposure: relevance to second-hand smoking, electronic cigarette use, and compulsive smoking. Front Psychiatry. 2013 Jun 4;4:41. doi: 10.3389/fpsyt.2013.00041. eCollection 2013. PMID 23761766
- [Background] Cohen LM, al'Absi M, Collins FL Jr. Salivary cortisol concentrations are associated with acute nicotine withdrawal. Addict Behav. 2004 Nov;29(8):1673-8. doi: 10.1016/j.addbeh.2004.02.059. PMID 15451136
- [Background] Cohrs S, Rodenbeck A, Riemann D, Szagun B, Jaehne A, Brinkmeyer J, Grunder G, Wienker T, Diaz-Lacava A, Mobascher A, Dahmen N, Thuerauf N, Kornhuber J, Kiefer F, Gallinat J, Wagner M, Kunz D, Grittner U, Winterer G. Impaired sleep quality and sleep duration in smokers-results from the German Multicenter Study on Nicotine Dependence. Addict Biol. 2014 May;19(3):486-96. doi: 10.1111/j.1369-1600.2012.00487.x. Epub 2012 Aug 23. PMID 22913370
- [Background] Colrain IM, Trinder J, Swan GE. The impact of smoking cessation on objective and subjective markers of sleep: review, synthesis, and recommendations. Nicotine Tob Res. 2004 Dec;6(6):913-25. doi: 10.1080/14622200412331324938. PMID 15801567
- [Background] Duskova M, Simunkova K, Hill M, Hruskovicova H, Hoskovcova P, Kralikova E, Starka L. Higher levels of salivary alpha-amylase predict failure of cessation efforts in male smokers. Physiol Res. 2010;59(5):765-771. doi: 10.33549/physiolres.931889. Epub 2010 Apr 20. PMID 20406037
- [Background] Elder GJ, Wetherell MA, Barclay NL, Ellis JG. The cortisol awakening response--applications and implications for sleep medicine. Sleep Med Rev. 2014 Jun;18(3):215-24. doi: 10.1016/j.smrv.2013.05.001. Epub 2013 Jul 5. PMID 23835138
- [Background] Fernandez-Mendoza J, Vela-Bueno A, Vgontzas AN, Olavarrieta-Bernardino S, Ramos-Platon MJ, Bixler EO, De la Cruz-Troca JJ. Nighttime sleep and daytime functioning correlates of the insomnia complaint in young adults. J Adolesc. 2009 Oct;32(5):1059-74. doi: 10.1016/j.adolescence.2009.03.005. Epub 2009 Mar 27. PMID 19328540
- [Background] Frederick SL, Reus VI, Ginsberg D, Hall SM, Munoz RF, Ellman G. Cortisol and response to dexamethasone as predictors of withdrawal distress and abstinence success in smokers. Biol Psychiatry. 1998 Apr 1;43(7):525-30. doi: 10.1016/S0006-3223(97)00423-X. PMID 9547932
- [Background] Granger DA. Children's salivary cortisol, internalising behavior problems, and family environment: Results from the Concordia Longitudinal Risk Project. International Journal Of Behavioral Development 22(4): 707-728, 1998.
- [Background] Hamidovic A, de Wit H. Sleep deprivation increases cigarette smoking. Pharmacol Biochem Behav. 2009 Sep;93(3):263-9. doi: 10.1016/j.pbb.2008.12.005. Epub 2008 Dec 16. PMID 19133287
- [Background] Hatsukami DK, Hughes JR, Pickens RW. Blood nicotine, smoke exposure and tobacco withdrawal symptoms. Addict Behav. 1985;10(4):413-7. doi: 10.1016/0306-4603(85)90038-3. PMID 4091074
- [Background] Hatsukami DK, Dahlgren L, Zimmerman R, Hughes JR. Symptoms of tobacco withdrawal from total cigarette cessation versus partial cigarette reduction. Psychopharmacology (Berl). 1988;94(2):242-7. doi: 10.1007/BF00176853. PMID 3127852
- [Background] Jaehne A, Unbehaun T, Feige B, Lutz UC, Batra A, Riemann D. How smoking affects sleep: a polysomnographical analysis. Sleep Med. 2012 Dec;13(10):1286-92. doi: 10.1016/j.sleep.2012.06.026. Epub 2012 Sep 28. PMID 23026505
- [Background] Jaehne A, Loessl B, Barkai Z, Riemann D, Hornyak M. Effects of nicotine on sleep during consumption, withdrawal and replacement therapy. Sleep Med Rev. 2009 Oct;13(5):363-77. doi: 10.1016/j.smrv.2008.12.003. Epub 2009 Apr 2. PMID 19345124
- [Background] Kaneita Y, Ohida T, Takemura S, Sone T, Suzuki K, Miyake T, Yokoyama E, Umeda T. Relation of smoking and drinking to sleep disturbance among Japanese pregnant women. Prev Med. 2005 Nov-Dec;41(5-6):877-82. doi: 10.1016/j.ypmed.2005.08.009. Epub 2005 Oct 24. PMID 16246406
- [Background] Kirschbaum C, Strasburger CJ, Langkrar J. Attenuated cortisol response to psychological stress but not to CRH or ergometry in young habitual smokers. Pharmacol Biochem Behav. 1993 Mar;44(3):527-31. doi: 10.1016/0091-3057(93)90162-m. PMID 8451256
- [Background] Koob GF, Volkow ND. Neurobiology of addiction: a neurocircuitry analysis. Lancet Psychiatry. 2016 Aug;3(8):760-773. doi: 10.1016/S2215-0366(16)00104-8. PMID 27475769
- [Background] Ma L, Chen YH, Chen H, Liu YY, Wang YX. The function of hypothalamus-pituitary-adrenal axis in children with ADHD. Brain Res. 2011 Jan 12;1368:159-62. doi: 10.1016/j.brainres.2010.10.045. Epub 2010 Nov 12. PMID 20971091
- [Background] Miller GE, Chen E, Zhou ES. If it goes up, must it come down? Chronic stress and the hypothalamic-pituitary-adrenocortical axis in humans. Psychol Bull. 2007 Jan;133(1):25-45. doi: 10.1037/0033-2909.133.1.25. PMID 17201569
- [Background] Moraes H, Deslandes A, Maciel-Pinheiro Pde T, Correa H, Laks J. Cortisol, DHEA, and depression in the elderly: the influence of physical capacity. Arq Neuropsiquiatr. 2016 Jun;74(6):456-61. doi: 10.1590/0004-282X20160059. PMID 27332070
- [Background] Moreno-Coutino A, Calderon-Ezquerro C, Drucker-Colin R. Long-term changes in sleep and depressive symptoms of smokers in abstinence. Nicotine Tob Res. 2007 Mar;9(3):389-96. doi: 10.1080/14622200701188901. PMID 17365770
- [Background] Nater UM, Rohleder N, Schlotz W, Ehlert U, Kirschbaum C. Determinants of the diurnal course of salivary alpha-amylase. Psychoneuroendocrinology. 2007 May;32(4):392-401. doi: 10.1016/j.psyneuen.2007.02.007. Epub 2007 Apr 5. PMID 17418498
- [Background] Newhouse PA, Sunderland T, Narang PK, Mellow AM, Fertig JB, Lawlor BA, Murphy DL. Neuroendocrine, physiologic, and behavioral responses following intravenous nicotine in nonsmoking healthy volunteers and in patients with Alzheimer's disease. Psychoneuroendocrinology. 1990;15(5-6):471-84. doi: 10.1016/0306-4530(90)90070-p. PMID 1966302
- [Background] Ohayon MM. Prevalence and correlates of nonrestorative sleep complaints. Arch Intern Med. 2005 Jan 10;165(1):35-41. doi: 10.1001/archinte.165.1.35. PMID 15642872
- [Background] Patten CA, Choi WS, Gillin JC, Pierce JP. Depressive symptoms and cigarette smoking predict development and persistence of sleep problems in US adolescents. Pediatrics. 2000 Aug;106(2):E23. doi: 10.1542/peds.106.2.e23. PMID 10920179
- [Background] Palmer CD, Harrison GA, Hiorns RW. Association between smoking and drinking and sleep duration. Ann Hum Biol. 1980 Mar-Apr;7(2):103-7. doi: 10.1080/03014468000004111. PMID 7425536
- [Background] Persico AM. Predictors of smoking cessation in a sample of Italian smokers. Int J Addict. 1992 Jun;27(6):683-95. doi: 10.3109/10826089209068760. PMID 1612820
- [Background] Phillips BA, Danner FJ. Cigarette smoking and sleep disturbance. Arch Intern Med. 1995 Apr 10;155(7):734-7. PMID 7695462
- [Background] Phillips B, Berry D, Schmitt F, Patel R, Cook Y. Sleep quality and pulmonary function in the healthy elderly. Chest. 1989 Jan;95(1):60-4. doi: 10.1378/chest.95.1.60. PMID 2909357
- [Background] Pillar G, Malhotra A, Lavie P. Post-traumatic stress disorder and sleep-what a nightmare! Sleep Med Rev. 2000 Apr;4(2):183-200. doi: 10.1053/smrv.1999.0095. PMID 12531165
- [Background] Prosise GL, Bonnet MH, Berry RB, Dickel MJ. Effects of abstinence from smoking on sleep and daytime sleepiness. Chest. 1994 Apr;105(4):1136-41. doi: 10.1378/chest.105.4.1136. PMID 8162739
- [Background] Richardson HN, Lee SY, O'Dell LE, Koob GF, Rivier CL. Alcohol self-administration acutely stimulates the hypothalamic-pituitary-adrenal axis, but alcohol dependence leads to a dampened neuroendocrine state. Eur J Neurosci. 2008 Oct;28(8):1641-53. doi: 10.1111/j.1460-9568.2008.06455.x. PMID 18979677
- [Background] Rohleder N, Kirschbaum C. The hypothalamic-pituitary-adrenal (HPA) axis in habitual smokers. Int J Psychophysiol. 2006 Mar;59(3):236-43. doi: 10.1016/j.ijpsycho.2005.10.012. Epub 2005 Dec 2. PMID 16325948
- [Background] Rohleder N, Nater UM, Wolf JM, Ehlert U, Kirschbaum C. Psychosocial stress-induced activation of salivary alpha-amylase: an indicator of sympathetic activity? Ann N Y Acad Sci. 2004 Dec;1032:258-63. doi: 10.1196/annals.1314.033. PMID 15677423
- [Background] Sadeh A, Alster J, Urbach D, Lavie, P. Actigraphically based automatic bedtime sleep-wake scoring: Validity and clinical applications. Journal of Ambulatory Monitoring 2(3): 209-216, 1989.
- [Background] Scharf SM, Maimon N, Simon-Tuval T, Bernhard-Scharf BJ, Reuveni H, Tarasiuk A. Sleep quality predicts quality of life in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2010 Dec 22;6:1-12. doi: 10.2147/COPD.S15666. PMID 21311688
- [Background] Simon-Tuval T, Scharf SM, Maimon N, Bernhard-Scharf BJ, Reuveni H, Tarasiuk A. Determinants of elevated healthcare utilization in patients with COPD. Respir Res. 2011 Jan 13;12(1):7. doi: 10.1186/1465-9921-12-7. PMID 21232087
- [Background] Steptoe A, Ussher M. Smoking, cortisol and nicotine. Int J Psychophysiol. 2006 Mar;59(3):228-35. doi: 10.1016/j.ijpsycho.2005.10.011. Epub 2005 Dec 6. PMID 16337291
- [Background] Taghizadeh N, Vonk JM, Boezen HM. Lifetime Smoking History and Cause-Specific Mortality in a Cohort Study with 43 Years of Follow-Up. PLoS One. 2016 Apr 7;11(4):e0153310. doi: 10.1371/journal.pone.0153310. eCollection 2016. PMID 27055053
- [Background] Tarasiuk A, Greenberg-Dotan S, Simon T, Tal A, Oksenberg A, Reuveni H. Low socioeconomic status is a risk factor for cardiovascular disease among adult obstructive sleep apnea syndrome patients requiring treatment. Chest. 2006 Sep;130(3):766-73. doi: 10.1378/chest.130.3.766. PMID 16963673
- [Background] Tarasiuk A, Greenberg-Dotan S, Brin YS, Simon T, Tal A, Reuveni H. Determinants affecting health-care utilization in obstructive sleep apnea syndrome patients. Chest. 2005 Sep;128(3):1310-4. doi: 10.1378/chest.128.3.1310. PMID 16162723
- [Background] Targovnik JH. Nicotine, corticotropin, and smoking withdrawal symptoms: literature review and implications for successful control of nicotine addiction. Clin Ther. 1989 Nov-Dec;11(6):846-53. PMID 2558798
- [Background] Vendruscolo LF, Barbier E, Schlosburg JE, Misra KK, Whitfield TW Jr, Logrip ML, Rivier C, Repunte-Canonigo V, Zorrilla EP, Sanna PP, Heilig M, Koob GF. Corticosteroid-dependent plasticity mediates compulsive alcohol drinking in rats. J Neurosci. 2012 May 30;32(22):7563-71. doi: 10.1523/JNEUROSCI.0069-12.2012. PMID 22649234
- [Background] Van Lenten SA, Doane LD. Examining multiple sleep behaviors and diurnal salivary cortisol and alpha-amylase: Within- and between-person associations. Psychoneuroendocrinology. 2016 Jun;68:100-10. doi: 10.1016/j.psyneuen.2016.02.017. Epub 2016 Feb 26. PMID 26963376
- [Background] Wetter DW, Carmack CL, Anderson CB, Moore CA, De Moor CA, Cinciripini PM, Hirshkowitz M. Tobacco withdrawal signs and symptoms among women with and without a history of depression. Exp Clin Psychopharmacol. 2000 Feb;8(1):88-96. doi: 10.1037//1064-1297.8.1.88. PMID 10743908
- [Background] Winternitz WW, Quillen D. Acute hormonal response to cigarette smoking. J Clin Pharmacol. 1977 Jul;17(7):389-97. doi: 10.1002/j.1552-4604.1977.tb04621.x. PMID 881471
- [Background] Won CH, Kryger M. Sleep in patients with restrictive lung disease. Clin Chest Med. 2014 Sep;35(3):505-12. doi: 10.1016/j.ccm.2014.06.006. Epub 2014 Jul 24. PMID 25156766
- [Background] Zaparoli JX, Galduroz JC. Treatment for tobacco smoking: a new alternative? Med Hypotheses. 2012 Dec;79(6):867-8. doi: 10.1016/j.mehy.2012.09.009. Epub 2012 Oct 6. PMID 23046856
- [Background] Zaniewska M, Przegalinski E, Filip M. Nicotine dependence - human and animal studies, current pharmacotherapies and future perspectives. Pharmacol Rep. 2009 Nov-Dec;61(6):957-65. doi: 10.1016/s1734-1140(09)70157-4. PMID 20081230
- [Background] Zhang L, Samet J, Caffo B, Punjabi NM. Cigarette smoking and nocturnal sleep architecture. Am J Epidemiol. 2006 Sep 15;164(6):529-37. doi: 10.1093/aje/kwj231. Epub 2006 Jul 7. PMID 16829553